CLINICAL TRIAL: NCT00528333
Title: A Phase IIB, Randomized, Double-Blinded, Placebo-Controlled Study of Low Dose Cytarabine and Lintuzumab Compared to Low Dose Cytarabine and Placebo in Patients 60 Years of Age and Older With Previously Untreated AML
Brief Title: A Study of Lintuzumab (SGN-33) in Combination With Low Dose Cytarabine in Patients 60+ Years With AML
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Seagen Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: SG033-0003
Record Dates: First submitted 2007-09-10; First posted 2007-09-12 (Estimated); Last update posted 2015-01-07 (Estimated); Status verified 2014-12

CONDITIONS: Acute Myeloid Leukemia
Keywords: Lintuzumab; Antigens, CD33; Antibodies, Monoclonal; Leukemia, Myeloid, Acute; Hematologic Diseases; Leukemia
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Hematologic Diseases; Leukemia | interventions — lintuzumab; Cytarabine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Lintuzumab plus low dose cytarabine
  Interventions: Drug: Lintuzumab (SGN-33); Drug: Low dose cytarabine
- 2 (Active Comparator): Placebo plus low dose cytarabine
  Interventions: Drug: Low dose cytarabine; Drug: Placebo

INTERVENTIONS:
Drug: Lintuzumab (SGN-33) — 600 mg IV on days 1, 8, 15 and 22 of cycle 1 and days 1 and 15 of each subsequent 28-day cycle up to a maximum of 12 cycles.
  Other Names: SGN-33
  Arms: 1
Drug: Low dose cytarabine — 20 mg SC twice a day on days 1-10 of each 28 day cycle up to a maximum of 12 cycles.
  Other Names: Ara-C, Cytosar
Drug: Placebo — IV administration on days 1, 8, 15, and 22 of cycle 1 and days 1 and 15 of each subsequent 28-day cycle up to a maximum of 12 cycles
  Arms: 2

SUMMARY:
The purpose of this study is to assess whether there is a survival benefit with lintuzumab given in combination with low dose cytarabine versus low dose cytarabine and placebo in patients with AML.

ELIGIBILITY:
Inclusion Criteria:

* Untreated AML that occurred de novo, after prior exposure to chemotherapy for a separate malignancy, or evolved from an antecedent hematologic disorder.
* After being informed of the potential benefits and risks of available treatment options, patients must have declined intensive chemotherapy for AML.
* At least 20% blasts in blood or marrow.
* Must have a minimum of 50% leukemic blasts that express CD33.
* ECOG performance status score of 0 to 2.
* WBC less than 30,000/µL

Exclusion Criteria:

* No known diagnosis of acute promyelocytic leukemia or chronic myeloid leukemia.
* No other active systemic malignancies treated with chemotherapy within the last 12 months.
* Must not have received previous chemotherapy (except hydroxyurea) for AML.
* Must not have significantly abnormal kidney or liver disease.
* Must not have known human immunodeficiency virus (HIV).

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 211 (Actual)
Dates: Start 2007-09; Primary Completion 2010-08 (Actual); Study Completion 2010-08 (Actual)

PRIMARY OUTCOMES:
Overall survival | 12 months

SECONDARY OUTCOMES:
Complete blood counts (CBC), Transfusion Requirements, Infections or Fevers of Unknown Origin Requiring Hospitalization or IV Antibiotics | 13 months

CONTACTS AND LOCATIONS:
Overall Officials: Eric Sievers, MD, Study Director — Seagen Inc.
Locations (20):
- United States (20):
  - Southern Cancer Center, Mobile, Alabama
  - Tower Cancer Research Foundation, Beverly Hills, California
  - Glendale Memorial Hospital, Glendale, California
  - Kenmar Research Institute, Los Angeles, California
  - University of California Los Angeles, Los Angeles, California
  - Bay Area Cancer Research Group, Pleasant Hill, California
  - University of Colorado Cancer Center, Aurora, Colorado
  - Lakeland Regional Cancer Center, Lakeland, Florida
  - H. Lee Moffitt Cancer Center & Research Institute, Tampa, Florida
  - Rush University Medical Center, Chicago, Illinois
  - Joliet Oncology-Hematology Associates, Joliet, Illinois
  - Michigan State University, Breslin Cancer Center, Lansing, Michigan
  - Billings Clinic Cancer Research, Billings, Montana
  - Northshore University Hospital, Monter Cancer Center, Lake Success, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Western Pennsylvania Cancer Institute, Pittsburgh, Pennsylvania
  - Cancer Centers of the Carolinas, Greenville, South Carolina
  - University of Texas, MD Anderson Cancer Center, Houston, Texas
  - Gunderson Clinic, La Crosse, Wisconsin

REFERENCES:
- [Result] Sekeres MA, Lancet JE, Wood BL, Grove LE, Sandalic L, Sievers EL, Jurcic JG. Randomized phase IIb study of low-dose cytarabine and lintuzumab versus low-dose cytarabine and placebo in older adults with untreated acute myeloid leukemia. Haematologica. 2013 Jan;98(1):119-28. doi: 10.3324/haematol.2012.066613. Epub 2012 Jul 16. PMID 22801961